CLINICAL TRIAL: NCT05511753
Title: The Effect of Acupuncture on Patients With Noise-induced Hearing Loss -- Randomized, Single-blinded, Controlled Prospective Clinical Trial
Brief Title: The Effect of Acupuncture on Patients With Noise-induced Hearing Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH110-REC1-240
Record Dates: First submitted 2022-08-16; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Electroacupuncture; Noise Induced Hearing Loss; Hearing Loss, Noise-Induced
MeSH Terms: conditions — Hearing Loss, Noise-Induced | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pure tone audiometry improving (Experimental): Pure tone audiometry: observe changes in hearing ability Evaluation time: Before acupuncture treatment, 2 weeks, 4 weeks, 6 weeks after treatment, and 2 weeks after acupuncture treatment, pure-tone audiometry was performed. The pure tone audiometry measures the hearing thresholds of 2KHz, 4KHz and 8KHz respectively.
  Interventions: Device: electroacupuncture

INTERVENTIONS:
Device: electroacupuncture — Insert stainless steel needles into the above acupoints and twist the needles to get qi. In addition, electroacupuncture stimulation (intensity 1mA, frequency 2Hz) was applied to connect the ipsilateral Yifeng and Wangu, and the ipsilateral Zhongzhu and Quchi.

SUMMARY:
In an era of advanced industry and commerce, working in a noisy environment is one of the most important risk factors for hearing damage, especially among young and middle-aged people. Although acupuncture has been widely used to treat otology-related diseases, such as tinnitus, dizziness, and sudden deafness, there are few studies on the effect of noise-induced hearing loss.

DETAILED DESCRIPTION:
Therefore, the purpose of this study is to investigate the effect of acupuncture on patients with noise-induced hearing loss. This study is designed as a randomized, single-blind, control prospective clinical trial. Eighty subjects with noise-induced hearing loss were included in the criteria and randomly divided into the acupuncture group and the control group as follows: 1) In the acupuncture group, in addition to the conventional treatment, acupuncture on both sides of Baihui (GV20), Dazhui (GV14), Yifeng (TE17), Wangu (GB12), Zhongzhu (TE3), Quchi (LI11), and connecting Yifeng and Wangu, and Zhongzhu and Quchi are given electroacupuncture stimulation (intensity of 1mA, frequency of 2Hz), 3 times a week, 15 minutes each time, continuous 6 weeks; 2) The control group was given conventional treatment only. The main assessment is the hearing changes of the pure tone hearing test, which measure the hearing thresholds of 2KHz, 4KHz, and 8KHz respectively; the secondary assessment is the change of the tinnitus handicap index score. The evaluation time includes before acupuncture treatment, 2 weeks, 4 weeks, 6 weeks after treatment, and 2 weeks after the end of acupuncture treatment.

The results of this study are expected to prove that acupuncture can improve noise-induced hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* pure tone audiometry diagnosed noise-induced hearing loss
* age: 20 - 65

Exclusion Criteria:

* major medical disease -- cancer, renal disease
* pregnancy or milk women
* anti-coagulation use
* pacemaker use
* allergy to needle
* denied accept inform consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
pure tone audiometry observe changes in hearing | Before acupuncture treatment, 2 weeks, 4 weeks, 6 weeks after treatment, and 2 weeks after acupuncture treatment
  The pure tone test measures the hearing thresholds of 2KHz, 4KHz and 8KHz respectively.